CLINICAL TRIAL: NCT04265313
Title: Validity and Reliability of the Turkish Version of the Neck Dissection Impairment Index
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Izmir Bakircay University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Kadirhan Ozdemir, PT, PhD., Head of Geriatric Rehabilitation Department, Izmir Bakircay University
Other Study IDs: 2018-145
Record Dates: First submitted 2020-02-08; First posted 2020-02-11 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Quality of Life; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head and Neck Cancer patients: Turkish patients diagnosed with Head and Neck Cancer
  Interventions: Other: Measurement of Quality of Life

INTERVENTIONS:
Other: Measurement of Quality of Life — Quality of life will be measured using The Neck Dissection Impairment Index, Modified Constant-Murley Score, Short Form-36 Health Survey version-2.0.

SUMMARY:
One of the long-term effects of neck dissection applied to patients with head and neck cancer is shoulder dysfunction, which directly affects the quality of life. Patients complain of different degrees of shoulder joint problems following neck dissection . Shoulder syndrome in these patients is characterized by a set of symptoms including shoulder pain, abduction limitation, and scapular winging.The aim of this study is to make the Turkish Neck validity, reliability and cultural adaptation of the "Neck Dissection Impairment Index".

DETAILED DESCRIPTION:
In the literature, there are many questionnaires aimed at patients with head and neck cancer, developed both specifically and specifically for this patient group, evaluating the quality of life. Regarding the shoulder problems experienced by these patients, there is only one item in the literature called "The University of Michegan Head and Neck QOL (UMHNQOL) questionnaire" that evaluates shoulder pain. Apart from this, there is no other questionnaire in the literature that may adversely affect the quality of life to neck dissection and question both neck and shoulder problems together. The Neck Dissection Impairment Index evaluates the shoulder-related quality of life in a more comprehensive and more detailed manner according to the UMHNQOL questionnaire. The Neck Dissection Impairment Index evaluates the components of shoulder related quality of life in a wide range after neck dissection. Because the type of age, weight, radiotherapy and neck dissection are the most important variables affecting quality of life, patients in the high-risk group (e.g. young individuals, patients who have received radiotherapy and modified radical neck dissection) evaluated with the Neck Dissection Impairment Questionnaire can benefit from an earlier and more intensive rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily accepting to participate in the study
* Patients whose native language is Turkish
* Patients or healthy individuals who have completed a minimum 11-month recovery period after selective or modified neck dissection

Exclusion Criteria:

* Having a pathological condition in the neck or shoulder that is not related to the treatments associated with head and neck cancer
* Cancer recurrence at the time of the evaluations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Turkish patients diagnosed with head and neck patients
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Neck Dissection Impairment Index | At baseline
  It consists of 10 items. Scoring is done according to the 5-point Likert scale. The patients answer the questions in the index as "1 = Not at all, 2 = A little, 3 = A moderate amount, 4 = Quite a bit, 5 = A lot". In order to standardize the obtained raw score over 100 points, the formula "(raw score-10) / 40] × 100" is used. This index evaluates the quality of life associated with neck and shoulder problems that occur in the long term after neck dissection [6].

SECONDARY OUTCOMES:
Modified Constant-Murley Score | At baseline
  It is a modified version of the Constant-Murley score used to evaluate pain, daily life activities, strength, and normal range of motion patency in various shoulder problems. In this test protocol, which is divided into four sub-scales, pain (15 points), daily life activities (20 points), strength (25 points) and normal range of motion (40 points) including flexion, external rotation, abduction and internal rotation movements are scored separately. 100 points in total are tried to be obtained. Pain and daily life activities sub scales in the test protocol will be filled by the patient. Evaluation of force and normal range of motion sub-scales will be done by a physiotherapist using a dynamometer and a goniometer, respectively [7]. Turkish version, validity, reliability and cultural adaptation of the modified Constant-Murley Score test protocol was performed by Celik et al. [10].
Short Form-36 Health Survey version-2.0 | At baseline
  It is a questionnaire version in which the instructions in the Short Form 36 (SF-36) questionnaire consisting of 36 questions are developed, the length of the questions are shortened, more familiar, more understandable and simpler words are used, easier to complete, faster to read and reducing the given answers. This questionnaire is a multi-item questionnaire which includes physical functions (10 items), social functions (2 items), role limitations caused by physical problems (3 items), mental health (5 items), energy / fitness (4 items), pain (2 items) and general health perception (5 items) [8]. The score of each item is coded, collected and converted into a scale from 0 to 100 [11]. The Turkish version, validity, reliability and cultural adaptation of the short form-36 Health Status Questionnaire-2.0 were made by Celik et al. [12].

CONTACTS AND LOCATIONS:
Locations (1):
- Kadirhan Ozdemir, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Sobol S, Jensen C, Sawyer W 2nd, Costiloe P, Thong N. Objective comparison of physical dysfunction after neck dissection. Am J Surg. 1985 Oct;150(4):503-9. doi: 10.1016/0002-9610(85)90164-3. PMID 4051117
- [Background] Soo KC, Guiloff RJ, Oh A, Della Rovere GQ, Westbury G. Innervation of the trapezius muscle: a study in patients undergoing neck dissections. Head Neck. 1990 Nov-Dec;12(6):488-95. doi: 10.1002/hed.2880120607. PMID 2258287
- [Background] Shone GR, Yardley MP. An audit into the incidence of handicap after unilateral radical neck dissection. J Laryngol Otol. 1991 Sep;105(9):760-2. doi: 10.1017/s0022215100117232. PMID 1833491
- [Background] Leipzig B, Suen JY, English JL, Barnes J, Hooper M. Functional evaluation of the spinal accessory nerve after neck dissection. Am J Surg. 1983 Oct;146(4):526-30. doi: 10.1016/0002-9610(83)90246-5. PMID 6625099
- [Background] NAHUM AM, MULLALLY W, MARMOR L. A syndrome resulting from radical neck dissection. Arch Otolaryngol. 1961 Oct;74:424-8. doi: 10.1001/archotol.1961.00740030433011. No abstract available. PMID 14477989
- [Background] Taylor RJ, Chepeha JC, Teknos TN, Bradford CR, Sharma PK, Terrell JE, Hogikyan ND, Wolf GT, Chepeha DB. Development and validation of the neck dissection impairment index: a quality of life measure. Arch Otolaryngol Head Neck Surg. 2002 Jan;128(1):44-9. doi: 10.1001/archotol.128.1.44. PMID 11784253
- [Background] Constant CR, Gerber C, Emery RJ, Sojbjerg JO, Gohlke F, Boileau P. A review of the Constant score: modifications and guidelines for its use. J Shoulder Elbow Surg. 2008 Mar-Apr;17(2):355-61. doi: 10.1016/j.jse.2007.06.022. Epub 2008 Jan 22. No abstract available. PMID 18218327
- [Background] Ware JE Jr. SF-36 health survey update. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3130-9. doi: 10.1097/00007632-200012150-00008. No abstract available. PMID 11124729
- [Background] Heutte N, Plisson L, Lange M, Prevost V, Babin E. Quality of life tools in head and neck oncology. Eur Ann Otorhinolaryngol Head Neck Dis. 2014 Feb;131(1):33-47. doi: 10.1016/j.anorl.2013.05.002. Epub 2013 Nov 28. PMID 24291153
- [Background] Celik D. Turkish version of the modified Constant-Murley score and standardized test protocol: reliability and validity. Acta Orthop Traumatol Turc. 2016;50(1):69-75. doi: 10.3944/AOTT.2016.14.0354. PMID 26854052
- [Background] Ware, J., M. Kosinski, and J. Dewey, How to score version 2 of the SF-36 health survey. Lincoln, RI: Quality Incorporated, 2000.
- [Background] Celik D, Coban O. Short Form Health Survey version-2.0 Turkish (SF-36v2) is an efficient outcome parameter in musculoskeletal research. Acta Orthop Traumatol Turc. 2016 Oct;50(5):558-561. doi: 10.1016/j.aott.2016.08.013. Epub 2016 Nov 17. PMID 27866914